CLINICAL TRIAL: NCT00817882
Title: Changing Perceptions of Work Ability in People With Low Back Pain: Feasibility Randomised Controlled Trial and Economic Evaluation.
Brief Title: Working Well With Back Pain (Feasibility RCT of Vocational Rehabilitation)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Arthritis Research UK (Other)
Responsible Party: Paul Cartledge, University of Nottingham
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 17891
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-11

CONDITIONS: Low Back Pain
Keywords: vocational; rehabilitation; work; ability; low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): individually targeted vocational rehabilitation
  Interventions: Other: individually targeted vocational rehabilitation
- 2 (Active Comparator): routine back pain rehabilitation
  Interventions: Other: routine back pain rehabilitation

INTERVENTIONS:
Other: individually targeted vocational rehabilitation — individually targeted vocational rehabilitation over 4 month period, maximum of 10 sessions, in addition to routine back pain rehabilitation.
  Maximum of 25 participants with low back pain
  Arms: 1
Other: routine back pain rehabilitation — routine back pain rehabilitation Maximum of 25 patients with low back pain
  Arms: 2

SUMMARY:
Back pain has a major impact on people's ability to work. Health professionals need to know how they can best use their limited resources to address the occupational needs of people with chronic low back pain. Vocational rehabilitation is the process that helps people with health problems to stay at, return to and remain at work. This study comprises the second phase of a three year study of back pain and vocational rehabilitation. The first phase gathered data from patient interviews and postal surveys of GPs and GP practice managers. These findings have been used to inform this second phase; a feasibility randomised controlled trial. The participants will be thirty employed people with back pain who have been offered an NHS rehabilitation programme, and who are concerned about their ability to work with low back pain. Those who consent will be randomised into two groups. One group will receive routine rehabilitation. The other will receive routine rehabilitation plus an individually tailored vocational intervention carried out by the researcher. Following the trial, individual interviews will be carried out with each of the participants by an independent researcher. An economic study will evaluate the possibility of measuring the cost-effectiveness of the intervention. The hypothesis is that an enhanced vocational intervention plus routine rehabilitation will be more effective in improving patients' work ability than routine rehabilitation alone.

ELIGIBILITY:
Inclusion Criteria:

* low back pain
* offered routine rehabilitation
* employed
* concern about work ability due to low back pain
* referral by GP in South Nottinghamshire

Exclusion Criteria:

* not fluent in English

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-05; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
work ability | prospective

SECONDARY OUTCOMES:
self-efficacy | prospective

CONTACTS AND LOCATIONS:
Overall Officials: Carol M Coole, MSc, Principal Investigator — University of Nottingham; Avril Drummond, PhD, Study Director — University of Nottingham; Paul J Watson, PhD, Study Director — University of Leicester
Locations (1):
- University of Nottingham, Nottingham, United Kingdom